CLINICAL TRIAL: NCT02638311
Title: Using Normal Volunteer Whole Blood or Plasma Samples to Establish the 99th Percentile Upper Reference Limit (URL) for the Meritas Troponin I Test
Brief Title: 99th Percentile Upper Reference Limit (URL) for the Meritas Troponin I Test
Status: Completed | Type: Observational
Sponsor: Trinity Biotech (Industry)
Responsible Party: Sponsor
Other Study IDs: CP7001_6URL
Record Dates: First submitted 2015-12-14; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA plasma samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective multicenter sample collection and testing study.

DETAILED DESCRIPTION:
Prospective multicenter sample collection and testing study. Approximately 750 apparently healthy subjects, including healthy subjects with stable co-morbidities, age, gender and ethnicity dispersed will be eligible for enrollment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 21 years of age at the time of enrollment in the study.
2. Subjects with no medications or no changes in their medications in the last 3 months.
3. Subjects with and without chronic stable morbidities (i.e., renal insufficiency, hypertension, diabetes, hypercholesterolemia, pulmonary disorders, coronary disease, musculoskeletal disorders, etc.).
4. Subjects able to understand and sign the informed consent and the patient questionnaire.

Exclusion Criteria:

1. Subjects with a history of heart failure and/or, having received treatment for heart failure.
2. Subject with renal failure.
3. Subjects with a history of unstable heart disease or angina complaints.
4. Subjects with any change in their medication in the last 3 months (diabetics may have small variations in glucose medications but may not have unstable disease, or have suffered a diabetic crisis in the last 6 months).
5. Any known acute infection in the last 30 days.
6. Marathon runners or extreme athletes.
7. Pregnant (self-reported).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females >21 years of age from diverse geographical locations and ethnicity-dispersed populations with an equal gender distribution
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
99th percentile for Troponin results determined from whole blood and plasma in apparetly healthy volunteer population | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jim Rock, Study Director — Trinity Biotech
Locations (3):
- United States (3):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical Research South, Charleston, South Carolina
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No